CLINICAL TRIAL: NCT04118634
Title: Evaluation of Performances of Biomarkers in Pulmonary Embolism
Brief Title: A Registry Study on Biomarkers of Pulmonary Embolism
Acronym: BIO-PE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: PE2019
Record Dates: First submitted 2019-09-26; First posted 2019-10-08 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2019-09

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Group with PE: The criteria for confirmation of PE are:
  PE on spiral computed tomography (CT) proximal deep vein thrombosis on ultrasound (US) thromboembolic events objectively confirmed during the follow up
- Group without PE: The criteria for exclusion of PE are:
  low or moderate clinical probability and D-dimer ELISA <0.50 µg/mL or <10xage in patients older than 50 years and negative follow up low and moderate clinical probability and negative CT and negative follow up high clinical probability and negative CT, US and follow up.

SUMMARY:
The purpose of the study is to evaluate the value of biomarkers in the diagnosis and risk stratification of patients with suspected pulmonary embolism.

DETAILED DESCRIPTION:
Management of patients with acute pulmonary embolism is a serious problem. The rapid and accurate diagnosis and risk stratification of these patients is an important unmet clinical need. The aim of the study is to evaluate the value of biomarkers, alone or in combination, in the diagnosis and risk stratification of patients with suspected pulmonary embolism presenting to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years that presents to an emergency department
* With suspected PE defined as new onset of or worsening of shortness of breath or chest pain

Exclusion Criteria:

* Hemodynamic instability
* Life expectancy less than 3 months
* First symptoms 15 day or more before inclusion
* Inability to the follow-up visits
* Therapeutic anticoagulation for any indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department with suspected PE
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2015-04-18 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve of biomarkers for the diagnosis of PE | 2 years
  The ROC curve will be built, the area under the curve will be calculated with its confidence interval.
PE related death | 7 days
  Number of PE related death

SECONDARY OUTCOMES:
Symptomatic recurrent venous thromboembolic events | 2 years
  Number of symptomatic recurrent venous thromboembolic event

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, PhD, Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided